CLINICAL TRIAL: NCT02808507
Title: Comparative Effectiveness/Implementation of TB Case Finding in Rural South Africa
Acronym: Kharitode TB
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins Bloomberg School of Public Health (Other)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH); Perinatal HIV Research Unit of the University of the Witswatersrand (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 15-0005; R01AI116787-02 (NIH)
Record Dates: First submitted 2016-06-01; First posted 2016-06-21 (Estimated); Results first posted 2022-12-02 (Actual); Last update posted 2024-09-05 (Actual); Status verified 2024-08

CONDITIONS: Tuberculosis
MeSH Terms: conditions — Tuberculosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Facility-based screening (Experimental): This strategy will be implemented at all clinics (n=28) within this arm for 18 months. Study staff will encourage providers at each of the clinics to screen all consenting patients attending the clinic, regardless of the original reason for clinic presentation. Upon presenting for care (e.g., while waiting for their healthcare provider), patients will be informed about the study and screened for cough of any duration, fever, weight loss, or night sweats. Participants who are symptomatic and provide a sputum specimen (according to the clinic standard of care) will be given a study flyer informing them that they may be contacted by study staff, and a brief summary of the study. Per standard of care, all sputum samples will be sent to the local National Health Laboratory Service laboratory for Xpert testing.
  Interventions: Other: Active TB case finding
- Contact screening (Experimental): This arm is comprised of two sub-arms:
  In the household contact screening sub-arm, a mobile field team visits the household of each consenting newly diagnosed pulmonary TB index case. Each visit consists of a household census, consent of all eligible household members for TB screening, administration of a brief questionnaire, sputum collection for testing with Xpert Mycobacterium tuberculosis (MTB)/rifampin (RIF) and the offer of HIV testing.
  In the incentive-based contact screening sub-arm, all consenting newly diagnosed active TB cases are provided with 10 coupons for free TB screening to give to close contacts. When a contact presents at clinic with a coupon, they and the index case each receive a small amount of money. If the contact is diagnosed with active TB and starts treatment, the index case receives an additional larger amount of money. Each contact receives a brief questionnaire, TB symptom screen, optional HIV testing, and sputum sample collection for Xpert MTB/RIF.
  Interventions: Other: Active TB case finding

INTERVENTIONS:
Other: Active TB case finding — Active TB case finding (ACF) refers to any number of strategies used to identify individuals with active TB disease, outside of passive case finding. In passive case finding, individuals with symptoms present at health centers for diagnosis. In active case finding, the health system makes an effort to identify TB cases before they present passively.

SUMMARY:
The purpose of this study is to compare three strategies for finding TB cases in a rural Sub-Saharan African setting: 1) Screening all attendees of primary care clinics for TB; 2) Conducting household contact investigations of newly diagnosed TB cases; 3) Providing incentives to newly diagnosed TB cases and their contacts to promote contact screening for TB. For each intervention, investigators will measure comparative effectiveness in terms of cases identified as well as the cost-effectiveness and feasibility of implementation.

ELIGIBILITY:
Inclusion Criteria:

Facility-based screening arm

* Age 0-99 years
* Informed consent provided (or assent plus parent/guardian consent)
* Attending any of the study 28 study clinics in the facility-based screening arm

Contact tracing arm- Index Case

* Age 0-99 years
* Informed consent provided (or assent plus parent/guardian consent)
* Newly diagnosed (last 2 months) with TB at any of the 28 study clinics in the contact tracing arm

Contact tracing arm- Household Contact

* Age 0-99 years
* Informed consent provided (or assent plus parent/guardian consent)
* Living in the same household as an enrolled Index case (see above)

Contact tracing arm- Non-household Close Contact

* Age 0-99 years
* Informed consent provided (or assent plus parent/guardian consent)
* Referred to the study as a close contact of an enrolled Index case (see above)

Exclusion Criteria (all arms):

* Unable to provide informed consent.

Ages: 0 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 4852 (Actual)
Dates: Start 2016-07-18 (Actual); Primary Completion 2018-01-17 (Actual); Study Completion 2020-01-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Dowdy, MD, PhD, Principal Investigator — Johns Hopkins Bloomberg School of Public Health
Locations (2):
- South Africa (2):
  - Vhembe health subdistrict, Louis Trichardt, Limpopo
  - Waterberg health subdistrict, Mokopane, Limpopo

REFERENCES:
- [Derived] Baik Y, Hanrahan CF, Mmolawa L, Nonyane BAS, Albaugh NW, Lebina L, Siwelana T, Martinson N, Dowdy DW. Conditional Cash Transfers to Incentivize Tuberculosis Screening: Description of a Novel Strategy for Contact Investigation in Rural South Africa. Clin Infect Dis. 2022 Mar 23;74(6):957-964. doi: 10.1093/cid/ciab601. PMID 34212181
- [Derived] Hanrahan CF, Nonyane BAS, Mmolawa L, West NS, Siwelana T, Lebina L, Martinson N, Dowdy DW. Contact tracing versus facility-based screening for active TB case finding in rural South Africa: A pragmatic cluster-randomized trial (Kharitode TB). PLoS Med. 2019 Apr 30;16(4):e1002796. doi: 10.1371/journal.pmed.1002796. eCollection 2019 Apr. PMID 31039165
- [Derived] Kerrigan D, West N, Tudor C, Hanrahan CF, Lebina L, Msandiwa R, Mmolawa L, Martinson N, Dowdy D. Improving active case finding for tuberculosis in South Africa: informing innovative implementation approaches in the context of the Kharitode trial through formative research. Health Res Policy Syst. 2017 May 30;15(1):42. doi: 10.1186/s12961-017-0206-8. PMID 28558737

RESULTS

PARTICIPANT FLOW:
Groups:
- Facility-based Screening Arm: This strategy will be implemented at all clinics (n=28) within this arm for 18 months. Study staff will encourage providers at each of the clinics to screen all consenting patients attending the clinic, regardless of the original reason for clinic presentation. Upon presenting for care (e.g., while waiting for their healthcare provider), patients will be informed about the study and screened for cough of any duration, fever, weight loss, or night sweats. Participants who are symptomatic and provide a sputum specimen (according to the clinic standard of care) will be given a study flyer informing them that they may be contacted by our study staff, and a brief summary of the study. Per standard of care, all sputum samples will be sent to the local National Health Laboratory Service laboratory for Xpert testing.
- Contact Tracing Household-based Sub-arm: This strategy will be implemented for 18 months at half of the clinics within the contact tracing arm (n=14) and, after a six-month washout period, for 18 months in the other half of the clinics in that arm (n = 14). All adults (and guardians for children) with newly diagnosed pulmonary TB will be approached for enrolment as described above. Consenting patients (estimated as 1,575 subjects) will be asked for a home address (with landmarks), mobile phone number, and convenient time for a household visit. A mobile field team consisting of a nurse and lay health worker (both research staff) will circulate between the 14 primary care clinics, with notifications of all new TB cases made from the clinic to the team by mobile phone. The field team will visit the household of each consenting index case within two weeks of notification; each visit will consist of a household census (including demographic data), consent of all eligible household members for questioning and TB screening, administration of a brief questionnaire (including symptomatology, self-reported HIV and TB history, care-seeking behavior, and acceptability of the intervention), and sputum collection for testing with Xpert MTB/RIF. Each participant will also be offered voluntary HIV counselling and testing. The team will make up to three visits to each household as needed in order to approach all household contacts for study enrolment.
- Contact Tracing Incentive-based Sub-arm: This strategy will be implemented in the opposite half of the clinics randomized to contact investigation. All adults (and guardians of children) with newly diagnosed active TB will be identified and approached for enrolment as described above. However, rather than a household visit, each consenting individual will be provided with a set of 10 coupons to give to household members and close contacts whom the index case believes may be at greatest risk. These coupons will contain instructions on how to come to the clinic for free TB screening (e.g., when the study team will be at each clinic), and will have an expiration date of 2 months from the time of initial TB diagnosis. When a contact presents at the clinic with the coupon, the contact will receive a small amount of money and a transport allowance based on the distance travelled to the clinic. If the contact is diagnosed with active TB and starts treatment, the contact will receive an additional larger amount of money. Study staff will document which index case the contact is linked to, and whether the contact is diagnosed with active TB. At the end of the 2 month period in which the coupons are valid the index will receive a grocery voucher for the total incentive earned (e.g., total amount for contact(s) who presented for screening + total amount for contact(s) diagnosed with active TB and starting treatment).
Period: Overall Study
Arm/Group | Facility-based Screening Arm | Contact Tracing Household-based Sub-arm | Contact Tracing Incentive-based Sub-arm
Started | 1929 | 1413 | 1510
Completed | 1929 | 1413 | 1510
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Facility-based Screening Arm | Contact Tracing Household-based Sub-arm | Contact Tracing Incentive-based Sub-arm | Total
Number analyzed (Participants) | 1929 | 1413 | 1510 | 4852
Age, Customized [Median (Inter-Quartile Range); unit: years]
  Age | 38 [28 to 49] | 39 [30 to 49] | 38 [29 to 48] | 38 [30 to 49]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 794 | 582 | 630 | 2006
  Male | 1135 | 831 | 880 | 2846
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  South Africa | 1929 | 1413 | 1510 | 4852
HIV status [Count of Participants; unit: Participants]
  HIV positive | 1161 | 797 | 902 | 2860
  HIV negative | 562 | 340 | 373 | 1275
  HIV status unknown | 205 | 274 | 235 | 714
  HIV status missing | 1 | 2 | 0 | 3

OUTCOME MEASURES:

1. Primary Outcome: Treatment Initiation Ratio in Facility Versus Contact Investigation Clinics
Description: The primary analysis was based on the facility- level rate ratio, and we first calculated an unadjusted ratio of the treatment initiation rates between the two arms and the corresponding 95% confidence interval (CI). We then adjusted for any residual confounding by district stratification and the historical annual number of people started on TB following a two-stage approach. The first step of this approach fits a Poisson regression to the facility-level counts and the district and historical volume covariates irrespective of study arm. The residuals ratios, calculated as the ratio of the observed over the expected counts, are then used in the second stage to estimate the between-arm rate ratio and the corresponding 95% CI.
Time Frame: 18 months
Population: The population for this outcome consists of a sub-group of the total study population (those enrolled during the intervention period of July 18,2015 - January 17, 2018). All participants from the facility-based screening arm are included (n=1929), and the participants of the contact screening arm (n=1726) are included (this is a combination from the household-based and incentive-based screening arms).
Measure: Count of Participants; unit: Participants
Groups:
- Contact Screening: This arm is comprised of two sub-arms:
  In the household contact screening sub-arm, a mobile field team visits the household of each consenting newly diagnosed pulmonary TB index case. Each visit consists of a household census, consent of all eligible household members for TB screening, administration of a brief questionnaire, sputum collection for testing with Xpert Mycobacterium tuberculosis (MTB)/rifampin (RIF) and the offer of HIV testing.
  In the incentive-based contact screening sub-arm, all consenting newly diagnosed active TB cases are provided with 10 coupons for free TB screening to give to close contacts. When a contact presents at clinic with a coupon, they and the index case each receive a small amount of money. If the contact is diagnosed with active TB and starts treatment, the index case receives an additional larger amount of money. Each contact receives a brief questionnaire, TB symptom screen, optional HIV testing, and sputum sample collection for Xpert MTB/RIF.
  Active TB case finding: Active TB case finding (ACF) refers to any number of strategies used to identify individuals with active TB disease, outside of passive case finding. In passive case finding, individuals with symptoms present at health centers for diagnosis. In active case finding, the health system makes an effort to identify TB cases before they present passively.
Arm/Group | Facility-based Screening | Contact Screening
Number analyzed (Participants) | 1929 | 1726
Participants | 1929 | 1726
Statistical Analysis 1: Comparison: Facility-based Screening vs Contact Screening; The primary analysis was based on the facility-level rate ratio. We first calculated an unadjusted ratio of the treatment initiation rates between the two arms and the corresponding 95% CI. We first fit a Poisson regression to the facility-level counts and the district and historical volume covariates. The residuals ratios, calculated as the ratio of the observed over the expected counts, were then used in the second stage to estimate the between-arm rate ratio and the corresponding 95% CI; Test type: Other; p = 0.73, See above comments; Treatment initiation ratio = 1.04, 95% CI 2-sided [0.80 to 1.3]

2. Primary Outcome: Comparative Treatment Initiation Ratio in the Incentive-based Versus Household-based Contact Investigation Arms
Description: The primary outcome of the study was the comparative number of people with incident TB diagnosed and started on treatment at study clinics in the two contact tracing arms, excluding the six-month washout period.
Time Frame: 36 months
Population: This analysis population includes all participants enrolled in the two contact tracing sub-arms during the total study period of 36 months. It excludes participants from the facility-based screening arm. A total of 2,923 patients were started on TB treatment during the study period: 1,413 in clinics allocated to household-based contact investigation and 1,510 in clinics allocated to incentive-based contact investigation.
Measure: Count of Participants; unit: Participants
Arm/Group | Contact Tracing Household-based Sub-arm | Contact Tracing Incentive-based Sub-arm
Number analyzed (Participants) | 1413 | 1510
Participants | 1413 | 1510
Statistical Analysis 1: Comparison: Contact Tracing Household-based Sub-arm vs Contact Tracing Incentive-based Sub-arm; The primary outcome of the study was the comparative number of people with incident TB diagnosed and started on treatment at study clinics during the two study periods, excluding the six-month washout period. The number of people starting treatment for incident TB was calculated by performing a review of paper and electronic medical records at each clinic on a quarterly basis during the study; Test type: Other; p = 0.68, Poisson regression; Treatment initiation ratio = 1.05, 95% CI 2-sided [0.97 to 1.13] — Adjusted for district, study phase and clinic random effect

3. Secondary Outcome: Comparative Number of Secondary TB Cases Identified in Incentive-based Versus Household-based Contact Tracing
Description: The pre-specified secondary study outcome was the number of Xpert-based TB diagnoses made among enrolled contacts ("secondary cases") by arm.
Time Frame: 36 months
Population: The number of TB contacts screened in each contact investigation arm.
Measure: Count of Participants; unit: Participants
Arm/Group | Contact Tracing Household-based Sub-arm | Contact Tracing Incentive-based Sub-arm
Number analyzed (Participants) | 1413 | 1510
Participants | 17 | 17
Statistical Analysis 1: Comparison: Contact Tracing Household-based Sub-arm vs Contact Tracing Incentive-based Sub-arm; Test type: Other; p = 0.80, Poisson regression — The pre-specified secondary study outcome was the number of Xpert-based TB diagnoses made among enrolled contacts ("secondary cases") by arm; Prevalence ratio = 1.0, 95% CI 2-sided [0.51 to 1.95] — Adjusted for study phase and district

4. Secondary Outcome: Total Cost of Household Contact Investigation Strategies
Description: This measure is the total cost of household contact investigation in both the household-based and incentive-based arms in 2018 United States dollar (USD) collected from the societal perspective (including both health systems and patient-level costs). As these are actual measured (not estimated) costs, no 95% confidence interval is reported.
Time Frame: 36 months
Population: This population includes all enrolled index participants with TB and their enrolled contacts, per arm.
Measure: Number; unit: 2018 US dollars
Arm/Group | Contact Tracing Household-based Sub-arm | Contact Tracing Incentive-based Sub-arm
Number analyzed (Participants) | 2664 | 2720
2018 US dollars | 48760 | 58070

5. Secondary Outcome: Estimated Costs Per Contact Person Screened in the Household-based and Incentive-based Contact Investigation Arms
Description: These are estimated costs in 2018 USD for the cost per contact person screened in each arm, collected from the societal perspective including health system and patient-level costs.
Time Frame: 36 months
Population: These populations include all contact persons enrolled into each arm.
Measure: Mean (95% Confidence Interval); unit: 2018 US dollars
Arm/Group | Contact Tracing Household-based Sub-arm | Contact Tracing Incentive-based Sub-arm
Number analyzed (Participants) | 1882 | 1940
2018 US dollars | 26.44 [15.17 to 102.28] | 29.93 [20.32 to 114.66]

6. Secondary Outcome: Cost Per Secondary Case of TB Identified Among Contacts, Per Arm
Description: Cost were measured in 2018 US dollars from the societal perspective, including both health systems and patient level costs. Total costs per arm were divided by the number of secondary TB cases identified among contacts in that arm.
Time Frame: 36 months
Population: Individuals included in this population were the total number of secondary TB cases identified among contacts enrolled in each arm.
Measure: Mean (95% Confidence Interval); unit: 2018 US dollars
Arm/Group | Contact Tracing Household-based Sub-arm | Contact Tracing Incentive-based Sub-arm
Number analyzed (Participants) | 17 | 17
2018 US dollars | 2927 [1680 to 11323] | 2416 [2319 to 13085]

7. Secondary Outcome: Incremental Cost-effectiveness Ratio
Description: (Total costs of incentive-based contact investigation-total costs of household-based contact investigation)/(effectiveness of incentive-based contact investigation-effectiveness of household-based contact investigation)
Time Frame: 36 months
Population: Though the difference in total costs by arm is positive, the difference in effectiveness by arm is zero, therefore we cannot calculate the incremental cost effectiveness ratio as it would require dividing by zero.
Groups:
- ICER Contact Investigation Population: This includes both arms of contact investigation (household-based and incentive-based) combined together into one group from which to calculate the incremental cost-effectiveness ratio
Arm/Group | ICER Contact Investigation Population
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: 36 months of study data collection, lasting from July 2016-January 2020.
Description: As our intervention is the implementation and observation of routine South African standard of care (intensified screening for TB at clinics and contact tracing of newly identified TB cases), we do not anticipate any medical adverse events which may occur as a result of this research study. Therefore, AEs (including SAEs) will not be recorded and reported for this study.
Arm/Group | Facility-based Screening Arm | Contact Tracing Household-based Sub-arm | Contact Tracing Incentive-based Sub-arm
All-Cause Mortality (participants affected / at risk) | 0/1929 | 0/1413 | 0/1510
Serious Adverse Events (participants affected / at risk) | 0/1929 | 0/1413 | 0/1510
Other Adverse Events (participants affected / at risk) | 0/1929 | 0/1413 | 0/1510

LIMITATIONS AND CAVEATS:
* Clinics were purposively chosen based on having larger historical TB patient volume; findings may not generalize to smaller, more remote clinics.
* Clinics and patients not blinded to allocation, so cannot rule out possibility of resultant bias.
* 1/3 of the index patients with TB whom we approached for enrollment refused or were unable to be enrolled, and cannot rule out that they may have differed in some way associated with TB incidence among their contacts from those able to be enrolled.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-07-31): https://cdn.clinicaltrials.gov/large-docs/07/NCT02808507/Prot_SAP_000.pdf